CLINICAL TRIAL: NCT07365748
Title: Evaluation of Bacterial Contamination and Antimicrobial Efficacy on Charcoal-Infused vs, Standard Nylon Toothbrush Bristles.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MTI University (Other)
Responsible Party: Principal Investigator, Esraa Hamed Aly, Lecturer of Pediatric Dentistry & Dental Public Health at MTI University, MTI University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SUEZ Med - IRB Approval No: 95
Record Dates: First submitted 2026-01-04; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: to Evaluate Antimicrobial Effect of Eco-friendly Toothbrush
Keywords: Eco-Friendly toothbrush , Charcoal toothbrush , Antimicrobial

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Antimicrobial effect of Eco-friendly tooth brush in children (Experimental): this arm will use the Eco-friendly toothbrush and will be evaluated for its antimicrobial effect
  Interventions: Device: Eco-friendly toothbrush for children
- Antimicrobial effect of Eco-friendly tooth brush in adults (Experimental): this arm will use the eco-friendly toothbrush and tested for its antimicrobial effect in adults
  Interventions: Device: Eco-friendly toothbrush in adults
- Nylon bristles toothbrush in children (Active Comparator): this arm will use the nylon toothbrush bristles and be evaluated for its antibacterial effect
  Interventions: Device: nylon bristles toothbrush in children
- nylon toothbrush bristles in adults (Active Comparator): this arm will use the nylon bristles toothbrush and be evaluated for its antimicrobial effect
  Interventions: Device: Nylon bristles toothbrush in adults

INTERVENTIONS:
Device: Eco-friendly toothbrush for children — it is an eco-friendly charcoal toothbrush assumed to have antibacterial property in children
  Arms: Antimicrobial effect of Eco-friendly tooth brush in children
Device: nylon bristles toothbrush in children — a normal man made toothbrush used by children
  Arms: Nylon bristles toothbrush in children
Device: Nylon bristles toothbrush in adults — a normal man made toothbrush used by adults
  Arms: nylon toothbrush bristles in adults
Device: Eco-friendly toothbrush in adults — to see the antimicrobial effect of eco-friendly toothbrush in adults
  Arms: Antimicrobial effect of Eco-friendly tooth brush in adults

SUMMARY:
This study compares two types of toothbrushes to see which one stays cleaner after use. Researchers want to know if toothbrushes with charcoal-infused bristles have fewer bacteria than standard toothbrushes with nylon bristles.

Participants in this study are adults and children who do not have gum disease or other major health issues. Everyone in the study will be assigned one of two types of toothbrushes:

* An eco-friendly toothbrush with charcoal bristles.
* A standard toothbrush with nylon bristles. Participants will use their assigned toothbrush at home for two specific time periods (one day and one week). They will follow simple instructions on how to brush and store the toothbrush. After each time period, they will return the toothbrush to the researchers.

The research team will test the bristles in a lab to count the bacteria. They will also measure how well the charcoal bristles stop bacteria from growing compared to the nylon bristles. This will help determine if charcoal toothbrushes are a more sanitary and eco-friendly option for daily oral care.

DETAILED DESCRIPTION:
Study Design and Randomization This study employs a randomized, parallel-group, ex-vivo microbiological design to assess bacterial retention and antimicrobial efficacy. Participants are stratified by age (children and adults) and randomized to receive either an eco-friendly charcoal-infused toothbrush or a standard nylon toothbrush. Allocation is managed using computer-generated random sequences concealed in sequentially numbered, opaque envelopes. To maintain blinding, laboratory outcome assessors are unaware of group assignment, and participants are instructed not to disclose their intervention to the assessment team.

Standardized Usage Protocol

To minimize variability in bacterial load due to behavioral factors, all participants adhere to a strict hygiene protocol:

* Brushing Technique: Participants brush twice daily (morning and evening) for two minutes using a standardized method (45-degree angle to the gingiva with short back-and-forth strokes, and vertical strokes for anterior lingual surfaces).
* Storage and Maintenance: Post-brushing, bristles are rinsed under running water without digital manipulation. Toothbrushes must be stored upright, uncovered, and positioned at least two feet away from sanitary fixtures (e.g., toilets) to minimize aerosol contamination.
* Restrictions: The use of antimicrobial mouthrinses, medicated toothpastes, or bristle covers is prohibited during the active study phases.

Sample Collection Timeline

The study involves two distinct usage periods separated by a washout phase:

1. Phase 1 (24-Hour Assessment): Participants use the assigned toothbrush for one day, followed by immediate return in a sterile pouch.
2. Washout: A 7-day period occurs where participants revert to their non-study oral hygiene routine.
3. Phase 2 (7-Day Assessment): Participants receive a new toothbrush of the same allocation, use it for 7 days, and return it in a sterile pouch for analysis.

Microbiological Analysis Returned samples are processed under aseptic laboratory conditions. Approximately one-third of the bristle field is excised using sterile instrumentation and transferred to test tubes containing 5 mL of sterile saline. The tubes are agitated to elute adherent microorganisms into suspension. A 0.1 mL aliquot is inoculated onto blood agar plates using a sterile spreader.

Plates are incubated in anaerobic gas pack jars at 37°C. Colony Forming Units (CFUs) are quantified after 48 hours of incubation to determine total bacterial load. Additionally, the intrinsic antimicrobial activity of the bristles is evaluated by measuring the zone of inhibition (in millimeters) surrounding bristle samples placed on agar plates after 7days of incubation.

ELIGIBILITY:
Inclusion Criteria:

* Participants free of any systemic diseases.
* Participants falling into one of two specific age groups:

A) Children aged 8 to 11 years.

B) Adults aged 18 to 35 years.

* Willingness to use the assigned toothbrush type (Eco-friendly charcoal or standard nylon).
* Ability to follow study instructions regarding brushing technique and storage.

Exclusion Criteria:

* Patients with open carious lesions.
* Participants with poor oral hygiene, defined as plaque index scores greater than 2.
* Participants with severe gingivitis, defined as gingival index score greater than 2.
* Current throat infections.
* Irregular brushing frequency (not brushing twice daily).
* Current use of mouthwash or antibacterial toothpastes.
* Current smokers.
* Medically compromised individuals.
* Unwillingness to use a charcoal Eco-friendly toothbrush.

Ages: 8 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2025-11-11 (Actual); Primary Completion 2025-12-20 (Actual); Study Completion 2026-01-01 (Actual)

PRIMARY OUTCOMES:
Colony-forming units (CFU) | 10 days
  Bacterial load will be quantified as CFU per milliliter (CFU/mL) from toothbrush bristles after 1 day and 1 week of use. One-third of the bristles will be aseptically cut, placed in 5 mL sterile saline, mixed to elute bacteria, then 0.1 mL will be plated onto blood agar. Plates will be incubated under anaerobic conditions for 48 hours, then colonies will be counted and recorded as CFU/mL.

CONTACTS AND LOCATIONS:
Locations (1):
- Dental clinic, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
age, gender
Supporting Information: ICF, CSR
Time Frame: october 2025 to october 2026